CLINICAL TRIAL: NCT04610372
Title: Moderate Versus Ultra Hypofractionation or Brachytherapy for PRimary OligoMetastatic Prostate Cancer Treatment
Brief Title: 5500/20 vs. SABR or Brachytherapy for PRimary OligoMetastatic Prostate Cancer Treatment (PROMPT)
Acronym: PROMPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, Professor of Radiation Oncology, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-01207
Record Dates: First submitted 2020-10-14; First posted 2020-10-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Prostate Cancer
Keywords: prostate adenocarcinoma; oligometastases; radiotherapy; hypofractionation; brachytherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: There is one standard arm (5500/20) and 3 alternative arms. The alternative arms are selected at the treating center. Thus, each randomization is 2-way, but with a 3:1 weighting so that the 4 treatment arms have equal numbers of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- standard (Active Comparator): External beam radiotherapy to deliver 5500 centiGray (cGy) in 20 fractions to the prostate over 4 weeks
  Interventions: Radiation: Hypofractionated external beam radiotherapy
- High dose rate brachytherapy (Experimental): A single fraction of 19 Gray (Gy) is delivered to the prostate under anesthesia as an out patient.
  Interventions: Radiation: High dose rate brachytherapy
- Permanent seed implant brachytherapy (Experimental): A single permanent implant of radioactive Iodine-125 seeds is performed under anesthesia as an out patient to deliver 125 Gy to the prostate
  Interventions: Radiation: Permanent seed implant
- Stereotactic body radiotherapy (Experimental): 36.25 Gy is delivered to the prostate in 5 fractions given either weekly or every second day, using a SABR technique.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated external beam radiotherapy — 5500 cGy/20 fractions delivered 5 days per week over 4 weeks
  Arms: standard
Radiation: High dose rate brachytherapy — A single fraction of 19 Gy is delivered from an automated afterloading Iridium-192 source via interstitial catheters placed under ultrasound guidance
  Arms: High dose rate brachytherapy
Radiation: Permanent seed implant — Iodine-125 radioactive seeds are implanted permanently in the prostate in a single procedure under transrectal ultrasound guidance
  Other Names: Low dose rate brachytherapy
  Arms: Permanent seed implant brachytherapy
Radiation: Stereotactic body radiotherapy — External radiation using SABR technology delivers 36.25 Gy to the prostate in 5 fractions given either once weekly for 5 weeks or every second day over 2 weeks.
  Other Names: SABR
  Arms: Stereotactic body radiotherapy

SUMMARY:
We will investigate whether ultrahypofractionation using stereotactic ablative radiotherapy (SABR) or brachytherapy is as well-tolerated as moderately hypofractionated external beam radiotherapy (EBRT) for treating the prostate in patients with oligometastatic prostate cancer. Secondary aims include assessment of progression-free survival (PFS) and overall survival (OS) as well as cost-effectiveness. We hypothesize that ultrahypofractionation will maintain favorable toxicity profiles and quality of life while achieving comparable or better efficacy, thereby providing a convenient and cost-effective alternative to moderately hypofractionated EBRT.

DETAILED DESCRIPTION:
Men newly diagnosed with low volume oligometastatic prostate cancer defined as fewer than 5 bone metastases and/or non regional lymph node involvement who agree to treatment of the primary cancer with radiation will be randomized between standard moderately hypofractionated external radiotherapy (5500 centiGray/20 fractions as per Stampede trial) and one of 3 alternatives: stereotactic body radiotherapy (SABR) to deliver 36 Gy/5 fractions, or low dose rate Iodine 125 permanent seed implant or a single high dose rate temporary implant. The trial will take place in 4 regional cancer centers of British Columbia Cancer Agency, with each center choosing their preferred alternative to 5500/20. To achieve 4 equally sized treatment arms, each randomization is weighted 3:1 for 42 patients in each arm and 168 total accrual. The primary endpoint is urinary quality of life as assessed by the International Prostate Symptom Score (IPSS) . As the typical acute symptoms from each of these radiation modalities has a unique time course, assessments are done at 6 different points during the first 2 years. Secondary endpoints are global quality of life as assessed by Expanded Prostate Cancer Index (EPIC) urinary, bowel and sexual scores, progression free survival, overall survival and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* European Cooperative Oncology Group performance status 0 to 2
* Medically fit for all protocol treatment and follow-up
* Histologically confirmed adenocarcinoma of the prostate
* Newly diagnosed any Tumor stage, any Nodal stage but with oligo metastases
* No prior therapy for prostate cancer apart from androgen deprivation
* Able to complete the necessary investigations prior to randomization (History and physical examination, PSA)
* Able to complete the necessary investigations prior to start of Radiotherapy (Transrectal ultrasound-guided biopsy or equivalent, CT chest, abdomen & pelvis or MRI abdomen and pelvis, and Bone scan)
* Planned for long-term androgen deprivation therapy (greater than 9 months in duration)
* Patient is able and willing to complete the quality of life questionnaires, and other assessments that are a part of this study

Exclusion Criteria:

* High metastatic burden defined as 5 or more bone metastases or visceral metastases
* Abnormal liver function
* Contraindications to EBRT such as active inflammatory bowel disease or previous pelvic radiation

Contraindications to brachytherapy including:

* Medically unfit for anesthesia,
* International Prostate Symptom Score (IPSS) greater than 20
* Poor urinary flow with peak flow rate less than10 mL per second or post-void residual greater than 25 per cent of voided volume (when uroflowmetry available)
* Prostate volume greater than 60cc after maximal cytoreduction
* Pubic arch interference
* Transurethral resection of prostate (TURP) within 12 weeks of brachytherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms | Baseline to 2 years
  International Prostate Symptom score (0/35), higher worse

SECONDARY OUTCOMES:
Expanded Prostate Cancer Index (EPIC) urinary domain | Baseline to 2 years
  Urinary Quality of life, 0/100 higher score better
EPIC bowel domain | Baseline to 2 years
  Bowel quality of life, 0/100, higher score better. Series of validated questions concerning urgency, frequency, consistency, leakage, presence of blood and pain with bowel movements and then rates how big a problem each symptom was (0-5)
EPIC sexual domain | Baseline to 2 years
  Sexual quality of life, 0/100, higher score better. Series of validated questions concerning frequency and quality of erections, presence of morning erections, ability to engage in sexual activity or intercourse, rates ability and then rates importance of each issue to the patient.
Biochemical failure (time to increase in prostate specific antigen (ng/ml) to 50% > nadir | Baseline to 3 years
  Progression free survival measured as time to Prostate Specific Antigen (PSA) rise by 50% > nadir
Distant metastatic failure | Baseline to 3 years
  Progression free survival measured as time to new or progressive bone metastases
Nodal progression | Baseline to 3 years
  Progression free survival measured as new or progressive adenopathy on imaging
Overall survival | 3 years
  Overall survival regardless of cause of death
Cause specific survival | Within 3 years of treatment
  Death from prostate cancer
Cost effectiveness | 3 years
  Analysis of primary treatment costs and secondary treatment costs at time of progression

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Crook, MD, Principal Investigator — BCCancer
Locations (4):
- Canada (4):
  - British Columbia Cancer Agency Center for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Center, Surrey, British Columbia
  - Vancouver Cancer Center, Vancouver, British Columbia
  - Vancouver Island Cancer Center, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No